CLINICAL TRIAL: NCT03515538
Title: A Phase 2a Randomized, Parallel Group, Open Label, Multicenter Study to Assess the Safety and Efficacy of RRx-001 in the Attenuation of Oral Mucositis in Patients Receiving Chemoradiation for the Treatment of Locally Advanced Squamous Cell Carcinoma of the Oral Cavity or Oropharynx
Brief Title: Safety and Efficacy of RRx-001 in the Attenuation of Oral Mucositis in Patients Receiving Chemoradiation for the Treatment of Oral Cancers
Acronym: PREVLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Collaborators: Prothex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR-001
Record Dates: First submitted 2018-04-18; First posted 2018-05-03 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Oral Mucositis
Keywords: head and neck cancer; squamous; neck cancer; oral cancer; mucositis; sores; mouth
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Mouth Neoplasms; Mucositis | interventions — RRx-001; Cisplatin; Injections; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RRx-001 Pre-Treatment plus SOC (Experimental): Two infusions of RRx-001 will be given each week during the two weeks prior to the start of RT/cisplatin SOC (four doses total). No additional RRx-001 will be given during the course of RT/cisplatin
  Interventions: Drug: RRx-001; Drug: Cisplatin for injection; Radiation: Radiation Therapy
- RRx-001 Pre-Treatment, 2 Concurrent Doses plus SOC (Experimental): Two infusions of RRx-001 will be given each week during the two weeks prior to the start of RT/cisplatin SOC. In addition, one dose of RRx-001 will be given on the last radiation day in each of weeks 2 and 5 during RT/cisplatin administration
  Interventions: Drug: RRx-001; Drug: Cisplatin for injection; Radiation: Radiation Therapy
- RRx-001 Pre-Treatment, 6 Concurrent Doses plus SOC (Experimental): Two infusions of RRx-001 will be given each week during the two weeks prior to the start of RT/cisplatin SOC. In addition, one dose of RRx-001 will be given on the last radiation day of each of the first 6 weeks during RT/cisplatin administration
  Interventions: Drug: RRx-001; Drug: Cisplatin for injection; Radiation: Radiation Therapy
- Standard of Care (Active Comparator): No doses of RRx-001 will be administered. Patients assigned to this arm will receive only standard of care in the form of a 7-week course of fractionated radiation therapy concurrent with a high-dose cisplatin regimen (100 mg/m2 dose in each of RT weeks 1, 4, and 7).
  Interventions: Drug: Cisplatin for injection; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: RRx-001 — RRx-001 for injection
  Arms: RRx-001 Pre-Treatment plus SOC; RRx-001 Pre-Treatment, 2 Concurrent Doses plus SOC; RRx-001 Pre-Treatment, 6 Concurrent Doses plus SOC
Drug: Cisplatin for injection — Patients will receive 3 doses of cisplatin at 100 mg/m2 in accordance with applicable guidelines such as NCCN; however, these guidelines are not intended to supersede or replace institutional guidelines with respect to appropriate and necessary care for individual patients
Radiation: Radiation Therapy — Intensity Modulated Radiation Therapy (IMRT) in accordance with the American College of Radiology (ACR) and American Society for Radiation Oncology (ASTRO) Practice Guideline for IMRT) is mandatory for this study

SUMMARY:
The purpose of this study is to determine if RRx-001, which is added on to the cisplatin and radiation treatment, reduces the duration or length of severe oral mucositis in patients with head and neck cancers. All patients in this study will receive 7 weeks of standard of care radiation therapy given with the chemotherapy agent, cisplatin. Patients in arms 1, 2 and 3 will also receive RRx-001 on different schedules.

DETAILED DESCRIPTION:
The standard treatment for head and neck cancer currently includes a chemotherapy drug called cisplatin that is given by intravenous (IV) infusion and radiation, which is delivered from a machine that precisely targets the tumor. One common and unfortunate side effect of treatment with cisplatin and radiation is oral mucositis, which refers to irritation of the lining of the mouth. Oral mucositis is a serious problem 1) because the open mouth sores from oral mucositis may lead to severe pain, nutritional problems and dehydration from an inability to eat and drink, an increased risk of infection from bacteria and fungus and delay or discontinuation of treatment and 2) because there is only one approved therapy to treat or prevent it.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of squamous cell carcinoma (SCC) of the oral cavity and oropharynx Note: Patients with unknown primary tumors whose treatment plan matches the requirements specified in Inclusion Criterion #3 below are eligible for the trial
2. Treatment planned to include standard cisplatin monotherapy administered either every three weeks (100 mg/m2 for 3 doses) with concomitant radiation delivered as a continuous course of IMRT with single daily fractions of 2.0 to 2.2 Gy with a cumulative radiation dose between 60 Gy and 72 Gy. Planned radiation treatment fields must include at least two oral sites (buccal mucosa, floor of mouth, tongue, soft palate) that are each planned to receive a total of > 55 Gy. Patients who have had prior surgery are eligible, provided they have fully recovered from surgery, and patients who may have surgery in the future are eligible.
3. ECOG performance status ≤ 2.
4. Participants must have adequate organ and marrow function as defined below:

   A. Absolute neutrophil count (ANC) >1,500 / mm3 B. Platelets > 100,000 / mm3 C. Hemoglobin ≥ 9.0 g/dL
5. Adequate renal and liver function as indicated by:

   A. Serum creatinine acceptable for treatment with cisplatin per institutional guidelines) B. Total bilirubin ≤ 1.5 x upper-normal limit (ULN) C. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN D. Alkaline phosphatase ≤ 2.5 x ULN
6. Human papilloma virus (HPV) status in tumor has been documented using tumor immunohistochemistry for HPV-p16 or other accepted test for patients with cancers of the oropharynx, base of tongue, or unknown primary.
7. Age 18 years or older
8. Patient must consent to the access, review and analysis of previous medical and cancer history, including imaging data by the sponsor or a third party nominated by the sponsor.
9. Ability to understand and sign a written informed consent document.
10. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

    Note: A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been postmenopausal for at least 12 consecutive months
11. Adequate visual access to permit examination of the following oral cavity sites: lips, buccal mucosa, floor of mouth, ventral and lateral tongue and soft palate.

Exclusion Criteria:

1. Prior radiation to the head and neck
2. Tumor of the lips, nasopharynx, hypopharynx, larynx, or salivary glands
3. Patients with simultaneous primaries or bilateral tumors
4. Metastatic disease (M1) Stage IV
5. Malignant tumors other than HNC within the last 5 years, unless treated definitively and with low risk of recurrence in the judgment of the treating investigator
6. Presence of oral mucositis (WHO Score ≥ Grade 1) or other oral mucosal ulceration at study entry
7. Grade 3 or 4 dysphagia or odynophagia (National Cancer Institute Common Toxicity Criteria, version 5.0) or inability to eat a normal diet
8. Requirement at baseline for parenteral or gastrointestinal tube-delivered nutrition for any reason
9. Known history of HIV or active hepatitis B/C (patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible)
10. Any significant medical diseases or conditions, as assessed by the investigators and sponsor that would substantially increase the medical risks of participating in this study (i.e., uncontrolled diabetes, NYHA II-IV congestive heart failure, myocardial infarction within 6 months of study, severe chronic pulmonary disease or active uncontrolled infection, uncontrolled or clinically relevant pulmonary edema).
11. Pregnant or nursing
12. Untreated active oral or dental infection, including severe tooth decay (caries)
13. Known allergies or intolerance to cisplatin and similar platinum-containing compounds
14. Evidence of immediate life-threatening disease or a life expectancy of less than 3 months
15. Receipt of unapproved or off-label medication within 30 days prior to start of study treatment
16. Sjogren syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, PhD, Study Director — EpicentRx, Inc.
Locations (12):
- United States (12):
  - John Wayne Cancer Institute @ Providence St. John's Health Center, Santa Monica, California
  - Centura Health Research Center, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Ballad Health, Johnson City, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
Started | 14 | 13 | 13 | 13
Completed | 9 | 10 | 9 | 8
Not Completed | 5 | 3 | 4 | 5
Not completed — Lack of Efficacy | 2 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Screen failure (baseline dropout) | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population comprises all subjects who are randomized and received at least 1 dose of study drug and will be used for all analyses of safety. Analysis is based on actual treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care | Total
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.17) | 56.7 (7.64) | 59 (11.94) | 59.5 (6.0) | 58.2 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 6
  Male | 10 | 9 | 12 | 9 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 11 | 10 | 13 | 9 | 43
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1 | 2
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 11 | 10 | 12 | 8 | 41
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 13 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Oral Mucositis (SOM)
Description: Duration in days of severe oral mucositis (SOM). Defined as oral mucositis grade 3 or 4 on the WHO Mucositis Grading Scale which comprises 5 grades: 0 = none, 1= oral soreness, erythema, 2 = oral erythema, ulcers, solid diet tolerated, 3 = oral ulcers, liquid diet only, and 4 = oral alimentation impossible. Severe Oral Mucositis duration is obtained by totaling the number of days a given patient experiences oral mucositis grade 3 or 4 during the randomized treatment period. Higher Severe Oral Mucositis duration numbers are indicative of worst outcomes. The total Severe Oral Mucositis duration for a given patient will range between 0 days and the maximum number of days the patient participated in the randomized treatment period.
Time Frame: From start of treatment through 28 days post treatment for up to 11 weeks from Start of Treatment
Population: All participants: number of days from the start of oral mucositis greater than a grade zero until resolution.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
Number analyzed (Participants) | 12 | 10 | 13 | 10
Days | 22.9 (19.08) | 27.7 (23.72) | 35.2 (28.83) | 37.8 (29.33)

2. Secondary Outcome: Time to Onset of Severe Oral Mucositis
Description: Time to onset of Severe Oral Mucositis defined as time (in days) from randomization to the first observed Severe Oral Mucositis. Longer Severe Oral Mucositis onset times are indicative of a better outcome. The time to onset of Severe Oral Mucositis for a given patient will range between 0 days and the maximum number of days the patient participated in the randomized treatment period.
Time Frame: Time from Day 1 to Oral Mucositis Onset (up to 8 weeks)
Population: All participants: number of days from start of treatment until participant experiences a OM grade of greater than zero.
Measure: Median (95% Confidence Interval); unit: Days to Onset
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
Number analyzed (Participants) | 12 | 10 | 13 | 10
Days to Onset | 38 [26 to NA] — insufficient number of participants with events | 33 [22 to NA] — insufficient number of participants with events | 37 [22 to NA] — insufficient number of participants with events | 26 [18 to NA] — insufficient number of participants with events

3. Secondary Outcome: Incidence of Severe Oral Mucositis
Description: Incidence of Severe Oral Mucositis defined as the number of patients who experienced a Severe Oral Mucositis grade 4 during the randomized treatment period.
Time Frame: Baseline through end of treatment (up to 11 weeks). Data collected every week.
Population: All participants who received study treatment and who experienced Oral Mucositis score greater than zero.
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
Number analyzed (Participants) | 12 | 10 | 13 | 10
Participants | 0 | 4 | 6 | 3

4. Secondary Outcome: Opioid Use
Description: Opioid use from the time to onset (TTO) and duration of opioid use among patients who were not taking opioids at radiation start or who required a second opioid during active treatment.
Time Frame: Baseline through end of radiation treatment (through 8 weeks). Data collected every week.
Population: Participants who required opioid use during treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
Number analyzed (Participants) | 12 | 10 | 13 | 9
Participants
  Week 1 | 1 | 0 | 0 | 1
  Week 2 | 2 | 0 | 1 | 2
  Week 3 | 4 | 2 | 2 | 4
  Week 4 | 4 | 2 | 2 | 4
  Week 5 | 4 | 2 | 3 | 4
  Week 6 | 4 | 2 | 3 | 4
  Week 7 | 4 | 2 | 3 | 4
  Week 8 | 4 | 2 | 4 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected beginning at baseline through end of treatment (12 weeks). All-Cause Mortality was assessed up to 12 weeks.
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 is used to grade adverse events.
Arm/Group | RRx-001 Pre-Treatment Plus SOC | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 1/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/12 | 4/11 | 6/13 | 5/10
Other Adverse Events (participants affected / at risk) | 9/12 | 10/11 | 12/13 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 Pre-Treatment Plus SOC (N=12) | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC (N=11) | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC (N=13) | Standard of Care (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001 Pre-Treatment Plus SOC (N=12) | RRx-001 Pre-Treatment, 2 Concurrent Doses Plus SOC (N=11) | RRx-001 Pre-Treatment, 6 Concurrent Doses Plus SOC (N=13) | Standard of Care (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 5 (8) | 4 (7) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 4 (4) | 2 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Flank pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Swelling face (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03515538/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03515538/ICF_001.pdf